CLINICAL TRIAL: NCT06033677
Title: "Intraoperative Use of Distal Radial Artery Cannulation With Snuffbox Approach'
Brief Title: Increasing Security With End-zone Arterial Blood Pressure Monitoring During Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Meral Erdal Erbatur, MD, Anesthesiology and reanimation spesialist, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 114-24/06/2022
Record Dates: First submitted 2023-08-22; First posted 2023-09-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Catheterization, Peripheral
Keywords: Invasive arterial pressure monitoring; Distal radial artery cannulation; Fovea radialis

STUDY DESIGN:
Intervention Model Description: Patients scheduled for elective surgery and requiring invasive arterial monitoring were divided into two groups.
  Group 1: The patients who were to undergo forearm radial artery catheterization were positioned with wrist dorsifection up to 30° and forearm supination. Intervention was planned after ultrasonographic measurements were taken.
  Group 2: The patients who will undergo distal radial artery catheterization were placed in the pronation position of the forearm with the anatomical snuffbox facing upwards. Intervention was planned after ultrasonographic measurements were taken.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grup 1-Forearm radial artery cannulation (FRA) (Other): The patients who were to undergo forearm radial artery catheterization were positioned with wrist dorsifection up to 30° and forearm supination. Intervention was planned after ultrasonographic measurements were taken.
  Interventions: Procedure: Forearm radial artery cannulation
- Grup 2-Distal radial artery cannulation (DRA) (Active Comparator): The patients who will undergo distal radial artery catheterization were placed in the pronation position of the forearm with the anatomical snuffbox facing upwards. Intervention was planned after ultrasonographic measurements were taken.
  Interventions: Procedure: Distal radial artery cannulation

INTERVENTIONS:
Procedure: Distal radial artery cannulation — Interventional application for invasive blood pressure monitoring
  Arms: Grup 2-Distal radial artery cannulation (DRA)
Procedure: Forearm radial artery cannulation — Interventional application for invasive blood pressure monitoring
  Arms: Grup 1-Forearm radial artery cannulation (FRA)

SUMMARY:
Short summary: The aim of this randomized controlled clinical research study was to compare distal radial artery cannulation with forearm radial artery cannulation in terms of efficacy and ease of administration. The investigators believe that cannulation of the distal radial artery in cases requiring invasive arterial monitoring should preserve the radial artery of the forearm for future health problems and reduce circulatory complications by working more distally.

The main question[s] aims to answer are:

* [question 1]: whether artery monitoring can be performed with a more distal approach
* [question 2]: efficacy and safety of the distal approach

DETAILED DESCRIPTION:
The distal radial artery (dRA) in the snuffbox location is a popular arterial access site for interventional cardiological procedures and neurointerventions. The investigators aimed to investigate the distal radial artery as an alternative site to the classical radial artery (RA) in cases requiring intraoperative arterial cannulation and blood pressure monitoring. The superficial location of the classic radial artery, its collateral blood flow with the ulnar artery, and limited complications make it a preferred choice for catheterization purposes. Given its use in various medical procedures such as flap transplantation, creating arteriovenous fistulas for hemodialysis, and bypass grafting, the investigators believe that preserving the classic radial artery is essential for potential health issues likely to arise in the future. In addition, the investigators aim to minimize circulatory complications by working more distally. Furthermore, it's worth mentioning that alterations in wrist positioning causing disruptions in the invasive arterial waveform also create a need for a different puncture approach. For all these conditions, the investigators believe that the snuffbox approach to distal radial artery cannulation would be an advantageous alternative.

This study will be a prospective randomized, controlled single-blind study. Patients who are scheduled for elective surgery, aged 18 and above, with ASA 1, 2, or 3 classifications, and requiring intraoperative arterial cannulation at Diyarbakır Gazi Yaşargil Training and Research Hospital will be included in the study. The exclusion criteria for participating in the study are as follows: under 18 years of age, ASA-4 classification, presence of non-palpable arteries, presence of burns or infection at the cannulation site, peripheral vascular disease, bleeding or coagulation disorders, negative modified Allen's test, and communication disorders. The withdrawal criteria for the study include a patient's desire to withdraw from the study at any stage and an extended cannulation time.

Participants will be divided into two groups, and ultrasound-guided cannulation will be performed for each group. One group will be cannulated through the classical radial artery of the forearm, while the other group will be cannulated through the distal radial artery using the snuffbox approach. Demographic data (age, gender, weight, height, BMI, comorbidity, medications, ASA, previous artery intervention, working position and working time), USG measurement data (diameter and depth of the artery) and procedural data (hand selection, first attempt success rate, arterial catheterization time, arterial posterior wall puncture rate, intraoperative artery waveform quality, postoperative compression time, and complications) will be recorded.

The sample size was determined by G-Power version 3.1.9.4, taking into account a two-tailed alpha error of 0.05, a power of 0.80, and an effect size of 0.5. Based on this savings and N2/N1 allocations of 0.98 in a previous study ( Distal radial artery as an alternative approach to forearm radial artery for perioperative blood pressure monitoring: a randomized, controlled, noninferiority trial Jingwei Xiong1 , Kangli Hui1 , Miaomiao Xu1 , Jiejie Zhou1 , Jie Zhang1 and Manlin Duan1,2* Xiong et al. BMC Anesthesiology (2022) 22:67 https://doi.org/10.1186/s12871-022-01609-5 ), the minimum number required for the study was planned to be 52 patients in the dRA group and 50 patients in the RA group.

The intervention will be performed under USG guidance by a single anesthesiologist with at least 5 years of experience in arterial cannulation.

The anticipated study duration is 6 months, and once approved by your institution, the study will commence and will be concluded upon reaching the target number of participants.

SPSS 21.0 for Windows software (SPSS Inc., Chicago, IL, USA) will be conducted for statistical analysis of the data. When evaluating the data statistically, numerical data will be expressed as mean and standard deviation, while categorical data will be presented as frequency and percentage. The chi-square test and Fisher's Exact test will be used to compare categorical data between groups, and the results will be reported as percentages (%n). Non-categorical data's normal distribution will be assessed using the Kolmogorov-Smirnov test. For normally distributed data, Student's t-test was used for statistical comparison between groups. For non-normally distributed data, the Mann-Whitney U test was employed. In all analyses, p-values less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for elective surgery
* Aged 18 and above
* ASA 1, 2, or 3 classifications
* Requiring intraoperative arterial cannulation
* At TC SBÜ Diyarbakır Gazi Yaşargil Training and Research Hospital will be included in the study

Exclusion Criteria:

* Under 18 years of age
* ASA-4 classification
* Presence of non-palpable arteries
* Presence of burns or infection at the cannulation site
* Peripheral vascular disease, bleeding or coagulation disorders
* Negative modified Allen's test, and communication disorders. The withdrawal criteria for the study include a patient's desire to withdraw from the study at any stage and an extended cannulation time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Number of interventions performed with USG guidance | during cannulation procedure
  The number of attempts will be recorded as 1st attempt, 2nd attempt and 3rd and above attempts.

SECONDARY OUTCOMES:
arterial catheterization time | during cannulation procedure
  Arterial catheterization time will be evaluated as under or over 3 minutes.
Monitored arterial waveform success | During the intraoperative period
  Monitored arterial waveform success will be evaluated as follows
  1. successful (there is a wave)
  2. fail (no wave)
  3. intraoperative damping time (the time during which the arterial wave disappears while the operation continues)
Compression time after catheter removal | procedure (the process until the catheter is removed and the bleeding stops)
  After the catheter is removed, the compression time will be measured in seconds. Bleeding will be checked every 30 seconds.
complication follow-up | Complication follow-up will be done from the beginning of cannulation procedure to the 24th hour postoperatively.
  Developing complications (vasospasm, hematoma, color and temperature change in the finger)
  1. During the intraoperative period,
  2. In the postoperative period
     * upon first arrival in the recovery room,
     * 1st hour at the end of the operation,
     * 6th hour at the end of the operation and
     * 24st at the end of the operation] will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Meral Edal Erbatur, M.D., Principal Investigator — University of Health Sciences Gazi Yasargil Training and Research Hospital
Locations (1):
- Health Sciences University Gazi Yaşargil Training and Research Hospital:, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamandi M, Saad M, Hasan R, Megaly M, Abbott JD, Dib C, Szerlip M, Potluri S, Lotfi A, Kiemeneij F, Al-Azizi KM. Distal Versus Conventional Transradial Artery Access for Coronary Angiography and Intervention: A Meta-Analysis. Cardiovasc Revasc Med. 2020 Oct;21(10):1209-1213. doi: 10.1016/j.carrev.2020.03.020. Epub 2020 Mar 14. PMID 32321695
- [Result] Hammami R, Zouari F, Ben Abdessalem MA, Sassi A, Ellouze T, Bahloul A, Mallek S, Triki F, Mahdhaoui A, Jeridi G, Abid L, Charfeddine S, Kammoun S, Jdidi J. Distal radial approach versus conventional radial approach: a comparative study of feasibility and safety. Libyan J Med. 2021 Dec;16(1):1830600. doi: 10.1080/19932820.2020.1830600. PMID 33147107